CLINICAL TRIAL: NCT01403545
Title: Safety, Tolerability and Pharmacokinetics of Liposomal Curcumin in Healthy Volunteers - A Phase I Dose Escalation Study
Brief Title: Evaluation of Liposomal Curcumin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SignPath Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Wolzt, M.D., Ao. Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lipocurc1001; 2011-001861-41 (EudraCT Number)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Drug Safety
Keywords: Safety; Tolerability; Pharmacokinetics; Liposomal Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Curcumin (Experimental): Single dose, dose escalation
  Interventions: Drug: Liposomal Curcumin
- 5% Glucose (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Liposomal Curcumin — Single dose intravenous infusion of liposomal Curcumin at 10, 20, 40, 80, 120, 180 mg/m² over 120 minutes
  Arms: Liposomal Curcumin
Other: Placebo — 5% glucose infusion over 120 minutes
  Arms: 5% Glucose

SUMMARY:
Aim of the present study is:

* To evaluate the safety and tolerability of increasing doses of intravenous liposomal Curcumin in healthy subjects by means of adverse events, vital signs and safety laboratory assessments.
* To investigate the pharmacokinetics of increasing doses of intravenous liposomal Curcumin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects.
* Age between 18-45 years.
* Body mass index between 18-27 kg/m2
* Vital signs within the normal range after 5 minutes in supine position (SBP: ≥90 mmHg and ≤140 mmHg, DBP: ≥45 mmHg and ≤90 mmHg, Heart rate: ≥45 bpm and ≤90 bpm).
* Normal ECG (PR-interval ≤ 210 ms, QRS duration ≤ 140 ms, QTc ≤ 450 ms).
* Adequate bone marrow function as evidenced by an absolute neutrophil count ≥1500 cells/µl, all normal red blood cell indices, hemoglobin greater than 11 g/dl and a platelet count greater than 150,000/µl.
* Normal renal function.
* Normal hepatic function as evidenced by serum total bilirubin ≤1.2 mg/dl, or less than or equal to the upper limit of normal, and alkaline phosphatase less than or equal to the upper limits of normal, and ASAT and ALAT less than or equal to the upper limits of normal.
* Normal coagulation profile, and activated partial thromboplastin time (aPTT).
* Normal urine analysis.
* Signed informed consent.

Exclusion Criteria:

* Intake of steroids within 2 weeks prior to the first dose of study drug.
* Concomitant medications (especially anticoagulants and aspirin) or herbal supplements.
* Active infection, or a fever > 38.5°C within three days prior to the first scheduled day of study drug dosing.
* Current or past history evidence of disease (e.g. hemolytic diathesis, anemia requiring substitution therapy, hemochromatosis) that could be exacerbated by administration of liposomal curcumin.
* History of prior malignancy within the past five years except for curatively treated non-melanoma skin cancer or cervical intraepithelial neoplasia.
* Allergy requiring medical treatment within the last four weeks.
* Known hypersensitivity to any of the components of turmeric.
* Participation in another clinical trial within 4 weeks before study initiation.
* NYHA Class 2 or congestive heart failure, uncontrolled hypertension, or arrhythmias.
* Positive HIV serology or evidence of active hepatitis.
* Unstable medical condition or any other medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with the patient's ability to sign the informed consent form, or his ability to cooperate and participate in the study, or to interfere with the interpretation of the results.
* History of treated or active seizure disorder or any CNS or PNS neurological disorder.
* Subjects who are pregnant or breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of increasing doses of intravenous liposomal Curcumin in healthy subjects by means of adverse events, vital signs and safety laboratory assessments. | From Baseline until 7 days after the study day

SECONDARY OUTCOMES:
Investigation of the pharmacokinetics of increasing doses of intravenous liposomal Curcumin in healthy subjects. | From Baseline until 48 hours after IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Storka A, Vcelar B, Klickovic U, Gouya G, Weisshaar S, Aschauer S, Bolger G, Helson L, Wolzt M. Safety, tolerability and pharmacokinetics of liposomal curcumin in healthy humans. Int J Clin Pharmacol Ther. 2015 Jan;53(1):54-65. doi: 10.5414/CP202076. PMID 25500488